CLINICAL TRIAL: NCT02009371
Title: A Clinical Study of Light Therapy on Depressive Episodes of Bipolar Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Xin Yu, President, Peking University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SF2011-4023-03
Record Dates: First submitted 2013-05-22; First posted 2013-12-12 (Estimated); Last update posted 2015-10-20 (Estimated); Status verified 2015-06

CONDITIONS: Depressive Episodes of Bipolar Disorder
MeSH Terms: interventions — Ultraviolet Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- Light therapy (Experimental): In this group, participants will be exposed to the LED treatment device (light box) which delivers bright light and meanwhile medicated with just one particular antipsychotics drug(a mood stabilizer or an atypical antipsychotic drug)except of antidepressants.
  Interventions: Device: Bright Light therapy
- Control group (Placebo Comparator): In this group, participants will be exposed to the same LED treatment device (light box) which delivers dim red light,which is considered to be biologically inactive, and meanwhile medicated with just one particular antipsychotics drug(a mood stabilizer or an atypical antipsychotic drug)except of antidepressants.
  Interventions: Device: dim Red Light therapy

INTERVENTIONS:
Device: Bright Light therapy — In this group, participants will be exposed to the LED treatment device (lightbox) which delivers bright light and meanwhile medicated with just one particular antipsychotics drug(a mood stabilizer or an atypical antipsychotic drug)except of antidepressants.
  Arms: Light therapy
Device: dim Red Light therapy — In this group, participants will be exposed to the same LED treatment device (light box) which delivers dim red light,which is considered to be biologically inactive, and meanwhile medicated with just one particular antipsychotics drug(a mood stabilizer or an atypical antipsychotic drug)except of antidepressants.
  Arms: Control group

SUMMARY:
The purpose of this study is to investigate the efficacy and safety of light-emitting diode(LED) light therapy on Chinese patients with Depressive Episodes of Bipolar Disorder and to gather prime research data and application parameters of LED light source which is not currently available in China.

ELIGIBILITY:
Inclusion Criteria:

* ages 18 to 65 years
* comply with the DSM-IV diagnosis of Bipolar I or II Disorder and a current depressive episode
* HAMD score ≥17 points
* intake of just one particular psychotropic drug(a mood stabilizer or an atypical antipsychotic drug) except of antidepressants and lasted 2 weeks.

Exclusion Criteria:

* inability to provide informed consent;
* previous treatment with BLT
* presence of another major psychiatric illness such as schizophrenia, schizoaffective disorder, lifetime alcohol or substance dependence
* diagnosed with a rapid-cycling bipolar disorder or currently in the mixed state or YMRS score>12 points
* use of antidepressants medications
* significant medical illness such as diabetes mellitus,heart failure, renal failure, severe liver function abnormalities,hyperthyroidism or hypothyroidism
* pregnancy;
* received magnified electroconvulsive therapy orRepetitive Transcranial Magnetic Stimulation in the past 3 months
* an eye condition that could be negatively affected by bright light
* suicidal risk or other factor making trial participation clinically inappropriate.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2013-01; Primary Completion 2015-03 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Reducing rate of HAMD | Change from baselin to 2 weeks after
  We used HAMD to evaluate the major state of depression.

SECONDARY OUTCOMES:
Reducing rate of CGI | Change from baseline to 2 week after
  We use CGI to evaluate the state of depression.

CONTACTS AND LOCATIONS:
Overall Officials: Xin Yu, professor, Principal Investigator — Peking University
Locations (1):
- Mental Health Institute of Peking University, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] LOOH,HALE A,D'HAENEN H. Detemination of the does of agomelatine,a melatoninergic agonist and selective 5-HT(2C) anlagonist,in the treatment of major depressive disorder:a placebo-controlled does range study[J].Int Clin Psychopharmacol,2002,17(5):239-247. OLIE JP,KASPER S. Efficacy of agomelatine,a MT1/MT2 receptor agonist with 5-HT(2C) antagonisitic properties, in major depressive disorder[J]. Int J Neuropsychopharmacol,2007,10(5):661-673. GUILLEMINAULT C. Efficacy of agomelatine versus venlafaxine on subjective sleep of patients with major depressive disorder [J]. Eur Neuropsychopharmacol,2005,15 Suppl3:S419-S420. LOPES MC.QUEPA-SALVAMA,GUILLEMINAULT C,Non-REM sleep instability in patinents with major depressive disorder;subjective improvement and improvement of non-REM sleep in stability with treatment(agomelatine)[J].Sleep Med,2007,9(1):33-41. Daniela Eser,Thomas C Baghai,etc.Agomelatine: The evidence for its place in the treatment of depression[J].Core Evidence 2009:3 171-179 Michele Fornaro, Davide Prestia,etc.A Systematic, Updated Review on the Antidepressant Agomelatine Focusing on its Melatonergic Modulation[J].Current Neuropharmacology, 2010, Vol. 8, No. 3:287-304 Chang-Ho Sohn,Raymond W. Lam.Update on the Biology of Seasonal Affective Disorder[J].CNS Spectr. 2005;10(8):635-646 Michael Terman,Jiuan Su Terman.Light Therapy for Seasonal and Nonseasonal Depression: Efficacy, Protocol, Safety, and Side Effects[J]CNS Spectr. 2005;10(8):647-663 Robert D. Levitan.Psychopharmacology for the Clinician Psychopharmacologie pratique[J].Rev Psychiatr Neurosci 2005;30(1)
- [Derived] Zhou TH, Dang WM, Ma YT, Hu CQ, Wang N, Zhang GY, Wang G, Shi C, Zhang H, Guo B, Zhou SZ, Feng L, Geng SX, Tong YZ, Tang GW, He ZK, Zhen L, Yu X. Clinical efficacy, onset time and safety of bright light therapy in acute bipolar depression as an adjunctive therapy: A randomized controlled trial. J Affect Disord. 2018 Feb;227:90-96. doi: 10.1016/j.jad.2017.09.038. Epub 2017 Sep 25. PMID 29053981